CLINICAL TRIAL: NCT01133340
Title: A Feasibility Study to Compare the Benefits of Endoscopic Tumor Clip Placement and 3T-MRI Simulation for Accurate Target Volume Definition for Rectal Cancer Patients Undergoing Pre-operative Chemoradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: IGAR Image guided adaptive radiotherapy (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECTAL MRI SIM 25409
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Rectal Cancer
Keywords: RADIOTHERAPY; CT simulation; MRI simulation; Endoscopic clip placement; Rectal cancer; Accuracy of MRI Simulation for target delineation and planning
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Radiation — No treatment intervention is planned. Patients will be scanned and treated as per department standards. The patient will have MRI at the time of their standard plan. They will then have clips inserted to mark the tumor after the standard scan is performed. The MRI and additional imaging with clips in place will be processed by 3 investigators who will contour based on the experimental image and compare this with the standard treated plan. Comparison of volumes in a blinded manner between investigators will also occur. The patients treatment will not be affected by the MRI or clip placement.

SUMMARY:
This study is looking for a better way to define rectal tumors undergoing pre-operative radiation. MRI scanning generally results in more clear definition of the tumor that CT scanning. Insertion of radio opaque clips in the tumor site could also help to visualize the tumor better for radiotherapy treatment planning. The investigators believe both techniques would help the physician to define to cancer better than using CT scan alone. The investigators also will compare both techniques to define the better way to define the tumor.

DETAILED DESCRIPTION:
1. The use of endoscopically placed mucosal metal clips to define the superior and inferior extent of the rectal tumor will improve the accuracy of tumor localization in patients undergoing non-contrast CT simulation.
2. A 3T-MRI will provide a better localization of the rectal tumor and pelvic nodes compared to non-contrast CT simulation for radiotherapy treatment planning.
3. By comparing these two novel methods to the standard procedure, we would be able to define any difference between the three methods and obtain an estimate of the accuracy and reliability of each method for the localization of the rectal tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the rectum stage as T3/4 N0/1/2 M0 undergoing pre-operative chemoradiation
* Patients must be 18 years of age or greater
* Signed study-specific informed consent
* Not pregnant or lactating

Exclusion Criteria:

* Contraindication for radiotherapy or chemoradiation
* Contraindication for MRI scanning
* Prior chemotherapy or radiation therapy to the pelvis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To define the usefulness of Endoscopic clip placement and 3T-MRI imaging for accurate target volume definition in rectal cancer patients undergoing pre-operative chemoradiation. | 1 year

SECONDARY OUTCOMES:
To assess the differences in pelvic lymph node (CTV) volume definition between Ct and MRI images. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kurian Joseph, MD, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada